CLINICAL TRIAL: NCT02777125
Title: A Randomized Trial Comparing Metered Dose Inhalers and Breath Actuated Nebulizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Mark Snider, Pediatric Emergency Medicine Fellow, Le Bonheur Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LeBonheurCH
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: pediatrics; metered dose inhalers; breath actuated nebulizers
MeSH Terms: conditions — Asthma | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol by Metered Dose Inhaler (Active Comparator): Albuterol administered via MDI and spacer device with weight and severity based dosing. For weight less than 20 kg: mild and moderate disease 540mcg of albuterol per dose. For weight greater than or equal to 20 kg: mild disease 540 mcg of albuterol per dose and moderate disease 1080 mcg of albuterol per dose.
  Interventions: Device: Metered Dose Inhaler
- Albuterol Breath Actuated Nebulizer (Active Comparator): Subjects randomized to BAN were evaluated for proper breath actuation technique. For subjects unable to coordinate breath actuation, the RT attached an appropriately sized mask to the device, changed the setting to continuous nebulization and returned upon completion of the treatment. Albuterol dosing was based upon the subject's weight and presenting symptom severity. Children presenting in the mild and moderate severity category weighing less than 20kg, received 2500mcg of albuterol. Children weighing more than 20kg, received 2500mcg of albuterol if their presentation met mild severity criteria, or 5000mcg if they met moderate criteria.
  Interventions: Device: Breath Actuated Nebulizer

INTERVENTIONS:
Device: Metered Dose Inhaler — A metered dose inhaler (MDI) is a small hand held pressurized canister device that contains both a medication, in this case albuterol, and a propellant. Pressing the device delivers 90mcg of albuterol. The MDI is attached to a spacer device, which is a one way holding chamber which allows the medication to be delivered over a series of breaths.
  Other Names: Aerochamber, AWA852-02
  Arms: Albuterol by Metered Dose Inhaler
Device: Breath Actuated Nebulizer — The breath actuated nebulizer (BAN) device is a device that converts liquid medication, in this case albuterol, into an aerosol. It consists of a mouthpiece, a medication reservoir, and connective tubing that attaches to a compressor. This BAN device delivers medication when the patient takes a breath, but it can be attached to a mask and set to continuous nebulization for patients that are not able to coordinate their breaths.
  Other Names: AeroEclipse
  Arms: Albuterol Breath Actuated Nebulizer

SUMMARY:
This study is determines if metered dose inhalers are as effective as breath actuated nebulizers for the treatment of mild to moderate asthma exacerbations in pediatric patients presenting to the emergency department. Half of the participating patients received albuterol via the metered dose inhaler whereas the other half received albuterol via the breath actuated nebulizer.

DETAILED DESCRIPTION:
Albuterol administered via metered dose inhalers with spacers are more effective than small volume nebulizers in the treatment of acute pediatric asthma exacerbations. There is also supporting data that the breath actuated nebulizers are also more effective than small volume nebulizers. The effectiveness of breath actuated nebulization compared to MDI for treating asthma exacerbations is less well defined.

Metered dose inhalers with spacers are more readily available to the general population, are easily transportable and do not require a power source. Demonstrating equal effectiveness of albuterol delivery systems for treatment of acute pediatric asthma exacerbations would enable physicians to confidently utilize clinical encounters as opportunities to educate families on management of asthma exacerbations using their home appliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting either with a first time wheeze or with an asthma exacerbation of a mild to moderate severity, both defined by a pediatric asthma score (PAS)11 of 5 to 11.

Exclusion Criteria:

* Subjects were excluded if they had initiated therapy at an outlying medical facility or had a history of any chronic lung disease
* Congenital heart disease, tracheostomy, or were receiving diuretic therapy.
* Patients diagnosed by the treating physician with bronchiolitis or pneumonia were excluded along with children who were wards of the state or whose parents did not speak English.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 980 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Snider, DO, Principal Investigator — University of Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naar-King S, Lam P, Ellis D, Bruzzese JM, Secord E. Asthma medication device skills in high-risk African American adolescents. J Asthma. 2013 Aug;50(6):579-82. doi: 10.3109/02770903.2013.786725. Epub 2013 May 28. PMID 23614823
- [Background] Reznik M, Silver EJ, Cao Y. Evaluation of MDI-spacer utilization and technique in caregivers of urban minority children with persistent asthma. J Asthma. 2014 Mar;51(2):149-54. doi: 10.3109/02770903.2013.854379. Epub 2013 Oct 22. PMID 24131031
- [Background] Reznik M, Jaramillo Y, Wylie-Rosett J. Demonstrating and assessing metered-dose inhaler-spacer technique: pediatric care providers' self-reported practices and perceived barriers. Clin Pediatr (Phila). 2014 Mar;53(3):270-6. doi: 10.1177/0009922813512521. Epub 2013 Dec 12. PMID 24336438
- [Background] Osmond MH, Gazarian M, Henry RL, Clifford TJ, Tetzlaff J; PERC Spacer Study Group. Barriers to metered-dose inhaler/spacer use in Canadian pediatric emergency departments: a national survey. Acad Emerg Med. 2007 Nov;14(11):1106-13. doi: 10.1197/j.aem.2007.05.009. Epub 2007 Aug 15. PMID 17699806
- [Background] Hussain-Rizvi A, Kunkov S, Crain EF. Does parental involvement in pediatric emergency department asthma treatment affect home management? J Asthma. 2009 Oct;46(8):792-5. PMID 19863282
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Amirav I, Newhouse MT. Metered-dose inhaler accessory devices in acute asthma: efficacy and comparison with nebulizers: a literature review. Arch Pediatr Adolesc Med. 1997 Sep;151(9):876-82. doi: 10.1001/archpedi.1997.02170460014003. PMID 9308864
- [Background] Leung K, Louca E, Coates AL. Comparison of breath-enhanced to breath-actuated nebulizers for rate, consistency, and efficiency. Chest. 2004 Nov;126(5):1619-27. doi: 10.1378/chest.126.5.1619. PMID 15539736
- [Background] Liu LL, Gallaher MM, Davis RL, Rutter CM, Lewis TC, Marcuse EK. Use of a respiratory clinical score among different providers. Pediatr Pulmonol. 2004 Mar;37(3):243-8. doi: 10.1002/ppul.10425. PMID 14966818
- [Background] Altamimi S, Robertson G, Jastaniah W, Davey A, Dehghani N, Chen R, Leung K, Colbourne M. Single-dose oral dexamethasone in the emergency management of children with exacerbations of mild to moderate asthma. Pediatr Emerg Care. 2006 Dec;22(12):786-93. doi: 10.1097/01.pec.0000248683.09895.08. PMID 17198210
- [Background] Chameides L, Ralston M, American Academy of Pediatrics, American Heart Association. Pediatric Advances Life Support. Dallas, Tx: American Heart Association;2011
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Sabato K, Ward P, Hawk W, Gildengorin V, Asselin JM. Randomized controlled trial of a breath-actuated nebulizer in pediatric asthma patients in the emergency department. Respir Care. 2011 Jun;56(6):761-70. doi: 10.4187/respcare.00142. Epub 2011 Feb 11. PMID 21333060
- [Background] Titus MO, Eady M, King L, Bowman CM. Effectiveness of a breath-actuated nebulizer device on asthma care in the pediatric emergency department. Clin Pediatr (Phila). 2012 Dec;51(12):1150-4. doi: 10.1177/0009922812458356. Epub 2012 Aug 28. PMID 22930778
- [Background] Arunthari V, Bruinsma RS, Lee AS, Johnson MM. A prospective, comparative trial of standard and breath-actuated nebulizer: efficacy, safety, and satisfaction. Respir Care. 2012 Aug;57(8):1242-7. doi: 10.4187/respcare.01450. Epub 2012 Feb 17. PMID 22348319
- [Background] Parone D, Stauss M, Reed CR, Sherman B, Smith L, Johnson R, Milcarek B, Hunter K. A comparative study of two nebulizers in the emergency department: breath-actuated nebulizer and handheld nebulizer. J Emerg Nurs. 2014 Mar;40(2):131-7. doi: 10.1016/j.jen.2012.10.006. Epub 2013 Jan 29. PMID 23369770
- [Background] Kerem E, Levison H, Schuh S, O'Brodovich H, Reisman J, Bentur L, Canny GJ. Efficacy of albuterol administered by nebulizer versus spacer device in children with acute asthma. J Pediatr. 1993 Aug;123(2):313-7. doi: 10.1016/s0022-3476(05)81710-x. PMID 8345434
- [Background] Ram FS, Wright J, Brocklebank D, White JE. Systematic review of clinical effectiveness of pressurised metered dose inhalers versus other hand held inhaler devices for delivering beta (2 )agonists bronchodilators in asthma. BMJ. 2001 Oct 20;323(7318):901-5. doi: 10.1136/bmj.323.7318.901. PMID 11668134
- [Background] Rodrigo C, Rodrigo G. Salbutamol treatment of acute severe asthma in the ED: MDI versus hand-held nebulizer. Am J Emerg Med. 1998 Nov;16(7):637-42. doi: 10.1016/s0735-6757(98)90164-4. PMID 9827736
- [Background] Doan Q, Shefrin A, Johnson D. Cost-effectiveness of metered-dose inhalers for asthma exacerbations in the pediatric emergency department. Pediatrics. 2011 May;127(5):e1105-11. doi: 10.1542/peds.2010-2963. Epub 2011 Apr 4. PMID 21464192
- [Background] Schuh S, Johnson DW, Stephens D, Callahan S, Winders P, Canny GJ. Comparison of albuterol delivered by a metered dose inhaler with spacer versus a nebulizer in children with mild acute asthma. J Pediatr. 1999 Jul;135(1):22-7. doi: 10.1016/s0022-3476(99)70322-7. PMID 10393599
- [Background] Leversha AM, Campanella SG, Aickin RP, Asher MI. Costs and effectiveness of spacer versus nebulizer in young children with moderate and severe acute asthma. J Pediatr. 2000 Apr;136(4):497-502. doi: 10.1016/s0022-3476(00)90013-1. PMID 10753248
- [Background] Rubilar L, Castro-Rodriguez JA, Girardi G. Randomized trial of salbutamol via metered-dose inhaler with spacer versus nebulizer for acute wheezing in children less than 2 years of age. Pediatr Pulmonol. 2000 Apr;29(4):264-9. doi: 10.1002/(sici)1099-0496(200004)29:43.0.co;2-s. PMID 10738013
- [Background] Castro-Rodriguez JA, Rodrigo GJ. beta-agonists through metered-dose inhaler with valved holding chamber versus nebulizer for acute exacerbation of wheezing or asthma in children under 5 years of age: a systematic review with meta-analysis. J Pediatr. 2004 Aug;145(2):172-7. doi: 10.1016/j.jpeds.2004.04.007. PMID 15289762
- [Background] Ploin D, Chapuis FR, Stamm D, Robert J, David L, Chatelain PG, Dutau G, Floret D. High-dose albuterol by metered-dose inhaler plus a spacer device versus nebulization in preschool children with recurrent wheezing: A double-blind, randomized equivalence trial. Pediatrics. 2000 Aug;106(2 Pt 1):311-7. doi: 10.1542/peds.106.2.311. PMID 10920157
- [Background] Staggs L, Peek M, Southard G, Gracely E, Baxendale S, Cross KP, Kim IK. Evaluating the length of stay and value of time in a pediatric emergency department with two models by comparing two different albuterol delivery systems. J Med Econ. 2012;15(4):704-11. doi: 10.3111/13696998.2012.674587. Epub 2012 Mar 23. PMID 22400716
- [Background] Zar HJ, Brown G, Donson H, Brathwaite N, Mann MD, Weinberg EG. Home-made spacers for bronchodilator therapy in children with acute asthma: a randomised trial. Lancet. 1999 Sep 18;354(9183):979-82. doi: 10.1016/s0140-6736(98)12445-5. PMID 10501359
- [Background] Zar HJ, Asmus MJ, Weinberg EG. A 500-ml plastic bottle: an effective spacer for children with asthma. Pediatr Allergy Immunol. 2002 Jun;13(3):217-22. doi: 10.1034/j.1399-3038.2002.01056.x. PMID 12144645
- [Background] Griffiths B, Ducharme FM. Combined inhaled anticholinergics and short-acting beta2-agonists for initial treatment of acute asthma in children. Cochrane Database Syst Rev. 2013 Aug 21;2013(8):CD000060. doi: 10.1002/14651858.CD000060.pub2. PMID 23966133
- [Background] Zorc JJ, Pusic MV, Ogborn CJ, Lebet R, Duggan AK. Ipratropium bromide added to asthma treatment in the pediatric emergency department. Pediatrics. 1999 Apr;103(4 Pt 1):748-52. doi: 10.1542/peds.103.4.748. PMID 10103297
- [Background] Goggin N, Macarthur C, Parkin PC. Randomized trial of the addition of ipratropium bromide to albuterol and corticosteroid therapy in children hospitalized because of an acute asthma exacerbation. Arch Pediatr Adolesc Med. 2001 Dec;155(12):1329-34. doi: 10.1001/archpedi.155.12.1329. PMID 11732951
- [Background] Wyatt EL, Borland ML, Doyle SK, Geelhoed GC. Metered-dose inhaler ipratropium bromide in moderate acute asthma in children: A single-blinded randomised controlled trial. J Paediatr Child Health. 2015 Feb;51(2):192-8. doi: 10.1111/jpc.12692. Epub 2014 Jul 14. PMID 25039574

RESULTS

PARTICIPANT FLOW:
Groups:
- Albuterol Breath Actuated Nebulizer: Subjects randomized to BAN were evaluated for proper breath actuation technique. The device settings were changed to provide continuous nebulization with a facemask if the patient could not breath actuate. Children presenting in the mild and moderate severity category weighing less than 20kg, received 2500mcg of albuterol. Children weighing more than 20kg, received 2500mcg of albuterol if their presentation met mild severity criteria, or 5000mcg if they met moderate criteria.
  Breath Actuated Nebulizer: The breath actuated nebulizer (BAN) device is a device that converts liquid medication, into an aerosol. It consists of a mouthpiece, a medication reservoir, and connective tubing that attaches to a compressor. This BAN device delivers medication when the patient takes a breath, but it can be attached to a mask and set to continuous nebulization for patients that are not able to coordinate their breaths.
Period: Overall Study
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Started | 488 | 492
Completed | 445 | 445
Not Completed | 43 | 47
Not completed — Consent form violation | 14 | 12
Not completed — Assent form violation | 21 | 23
Not completed — Protocol Violation | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer | Total
Number analyzed (Participants) | 445 | 445 | 890
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 445 | 445 | 890
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.37 (3.9) | 6.38 (4.0) | 6.37 (3.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 147 | 313
  Male | 279 | 298 | 577
Region of Enrollment [Number; unit: participants]
  United States | 445 | 445 | 890
Pediatric Asthma Score at Presentation [Mean (Standard Deviation); unit: units on a scale] — The Pediatric Asthma Severity Score is a composite score based upon the patient's respiratory rate, oxygen saturation, retractions, work of breathing and findings on auscultation. The score ranges from 5-15, with the higher score being associated with a more severe asthma exacerbation. A mild score ranges from 5-7, a moderate score of 8-11. The minimum score obtainable is 5, the maximum score is a 15. Any subject with a presenting score above 11 was not eligible for participation in this study as these would be classified as a severe exacerbation.
  units on a scale | 7.7 (1.7) | 8.0 (1.6) | 7.9 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant's Admitted to the Hospital for Further Treatment
Description: Patient disposition is measured as subjects requiring further treatment and being admitted to hospital. We record the number of patients in each cohort that required admission to the hospital after being evaluated and treated in the Emergency Department.
Time Frame: 6 hours
Measure: Number; unit: Participants admitted to the Hospital
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Number analyzed (Participants) | 445 | 445
Participants admitted to the Hospital | 53 | 57

2. Secondary Outcome: Emergency Department Length of Stay
Description: Emergency department length of stay is defined as the point of time when the patient checked into the Emergency Department to the time of final disposition.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Albuterol Breath Actuated Nebulizer: Subjects randomized to BAN were evaluated for proper breath actuation technique. For subjects unable to breath actuate, the RT changed the device setting to continuous nebulization, provided an appropriately sized mask, and returned upon completion of the treatment. Albuterol dosing was based upon the subject's weight and presenting symptom severity. Children presenting in the mild and moderate severity category weighing less than 20kg, received 2500mcg of albuterol. Children weighing more than 20kg, received 2500mcg of albuterol if their presentation met mild severity criteria, or 5000mcg if they met moderate criteria.
  Breath Actuated Nebulizer: The breath actuated nebulizer (BAN) device is a device that converts liquid medication, in this case albuterol, into an aerosol. It consists of a mouthpiece, a medication reservoir, and connective tubing that attaches to a compressor. This BAN device delivers medication when the patient takes a breath, but it can be atta
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Number analyzed (Participants) | 445 | 445
minutes
  Mild severity | 192 (96) | 197 (90)
  Moderate severity | 232 (125) | 245 (98)

3. Secondary Outcome: Number of Patients With Tachycardia After Treatment
Description: Defined as anytime after initiation of therapy when the patient's heart rate exceeded age adjusted normal sinus rhythm heart rates for their age. Not uncommonly, patient's experience tachycardia as an unintended side effect of receiving albuterol. Tachycardia can result in a patient requiring further observation in the Emergency department and therefore increasing Emergency Department length of stay. We want to determine if indeed tachycardia is unavoidable, or if its presence suggests that patients are receiving too much albuterol or if albuterol is being given by the wrong appliance.
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Number analyzed (Participants) | 445 | 445
Participants | 101 | 141

4. Secondary Outcome: Number of Patients Requiring Ondansetron Dosing
Description: Defined as a patient needing ondansetron for symptomatic relief of their nausea after initiating therapy in the Emergency Department.
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Number analyzed (Participants) | 445 | 445
Participants | 14 | 18

5. Secondary Outcome: Number of Participants Requiring Repeat Visits
Description: Defined as a repeat visit to the Emergency Department for a complaint related to their wheezing, within 7 days of initial enrollment in the study.
Time Frame: Within 7 days of initial presentation
Measure: Count of Participants; unit: Participants
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
Number analyzed (Participants) | 445 | 445
Participants | 5 | 4

ADVERSE EVENTS:
Groups:
- Albuterol Breath Actuated Nebulizer: Subjects randomized to BAN were evaluated for proper breath actuation technique. For subjects unable to breath actuate, the RT attached an appropriately sized mask to the device, changed the setting to continuous nebulization and returned upon completion of the treatment. Albuterol dosing was based upon the subject's weight and presenting symptom severity. Children presenting in the mild and moderate severity category weighing less than 20kg, received 2500mcg of albuterol. Children weighing more than 20kg, received 2500mcg of albuterol if their presentation met mild severity criteria, or 5000mcg if they met moderate criteria.
  Breath Actuated Nebulizer: The breath actuated nebulizer (BAN) device is a device that converts liquid medication, in this case albuterol, into an aerosol. It consists of a mouthpiece, a medication reservoir, and connective tubing that attaches to a compressor. This BAN device delivers medication when the patient takes a breath, but it can be atta
Arm/Group | Albuterol by Metered Dose Inhaler | Albuterol Breath Actuated Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/445 | 0/445
Serious Adverse Events (participants affected / at risk) | 0/445 | 0/445
Other Adverse Events (participants affected / at risk) | 101/445 | 141/445
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol by Metered Dose Inhaler (N=445) | Albuterol Breath Actuated Nebulizer (N=445)
Tachycardia (Cardiac disorders) | 101 (101) | 141 (141) — Incidence of age adjusted tachycardia prior to final disposition after receiving albuterol as per their randomized cohort according to our standard emergency department protocol

LIMITATIONS AND CAVEATS:
Unblinded study, eligible subjects may have been overlooked for fear of treatment failure. Recheck times were not standardized possibly affecting EDLOS and tachycardia. Baseline acuity differences between cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No